CLINICAL TRIAL: NCT00164697
Title: Legacy for Children, The CDC Parenting Research Projects
Brief Title: Legacy for Children, an Early Intervention Study to Promote Optimal Child Development in Low-income Families
Acronym: Legacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: RTI International (Other); University of California, Los Angeles (Other); University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDC-NCBDDD-2524; 200-94-0828; 200-98-0110; 200-98-0111
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2012-09

CONDITIONS: Child Development
Keywords: Child Development; Parenting; Child Rearing; Parent-Child Relations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Parenting group
  Interventions: Behavioral: Parenting group
- 2 (No Intervention): Families in this "usual care" comparison group were not prevented from utilizing any service that would otherwise be available to them, even if the service was similar to the services received in the intervention arm of the study.

INTERVENTIONS:
Behavioral: Parenting group — Weekly and periodic (10 weeks blocks with 6 week break) parenting group meetings (2.5-3 hr), periodic one-on-one meetings (2 hr), visits to community resources (2-3 hr per event). Legacy intervention activities are designed to enhance sensitive and responsive parenting, parent/child interaction, and promote a sense of community. Other activities include verbal and cognitive stimulation through parent and parent/child group meetings, visits to the home, and participation in community events.
  Other Names: Behavioral
  Arms: 1

SUMMARY:
The purpose of this study is to determine if an intervention focused on promoting parent-child interaction, parental responsibility, parental commitment of time and energy, and sense of community results in better developmental outcomes for low-income children.

DETAILED DESCRIPTION:
The early years of life (birth to age 5 years) are crucial in a child's development. Parents play a critical role in their children's development and are responsible for the environment in which they grow up. Past research shows that the personal characteristics of successful children consistently correlate to parental influences and behavior. Thus, the theoretical foundation in the Legacy study is that parents can positively influence their child's development. Also, parents are more likely to maintain positive parenting behaviors if they are part of a community greater than themselves. Legacy intervention activities are designed to enhance sensitive and responsive parenting, parent/child interaction, and promote a sense of community. Other activities include verbal and cognitive stimulation through parent and parent/child group meetings, visits to the home, and participation in community events. Legacy has both a pilot phase and a main study phase. There are 180 intervention and 120 comparison families in the main study phase and 60 of each in the pilot phase at each study site, Miami and Los Angeles. The 720 participating families are those whose children, on average, would be expected to fall below national norms on a range of developmental outcomes. Process, cost, and short- and long-term outcome data are being collected.

Comparison group: In addition to the current standard of care, the comparison families receive regular comprehensive child development and maternal assessments at 6 months, 1 yr, 2 yr, 3 yr, 4 yr, and 5 yr.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Live within 10 miles of UCLA
* 18 years of age or older
* Receive their prenatal and well-baby care from MediCal
* Live within 50 minutes of the three community intervention sites
* Reside within zip codes corresponding to the lowest performing schools in the broad Miami area
* Give birth to the target child at participating hospitals

Exclusion Criteria:

* Multiple birth greater than twins
* Existing Substance abuse
* Existing Mental Health issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 1999-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
child behavior | 1yr, 2 yr, 3 yr, 4 yr, 5 yr
child social skills | 1yr, 2 yr, 3 yr, 4 yr, 5 yr
child cognition | 1 yr, 3 yr, 5 yr
child language/communication | 2 yr, 4 yr, 5 yr
child attachment | 2 yr
child peer relationships | 5 yr
child academics | 4 yr, 5 yr
parent-child interaction | 6 months, 5 yr

SECONDARY OUTCOMES:
child physical growth | baseline, 6 month, 1 yr, 2 yr
child violence exposure | 2 yr, 4 yr, 5 yr
parenting | baseline, 6 mos, 2 yr, 3 yr 5 yr
maternal health | baseline, 1 yr 3 yr, 5 yr
maternal mental health | baseline, 1yr, 2yr, 3yr, 4 yr, 5 yr
sense of community | baseline, 1yr, 2yr, 3yr, 4 yr, 5 yr
community involvement | baseline, 6 mos, 2yr, 3yr, 5 yr
coping | 6mos, 2yr, 3 yr, 5 yr
HOME environment | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Perou, PhD, Principal Investigator — Centers for Disease Control and Prevention
Locations (2):
- United States (2):
  - UCLA Department of Pediatrics, Los Angeles, California
  - University of Miami School of Medicine, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barry CM, Robinson LR, Kaminski JW, Danielson ML, Jones CL, Lang DL. Behavioral and Socioemotional Outcomes of the Legacy for Children Randomized Control Trial to Promote Healthy Development of Children Living in Poverty, 4 to 6 Years Postintervention. J Dev Behav Pediatr. 2022 Jan 1;43(1):e39-e47. doi: 10.1097/DBP.0000000000000962. PMID 33941737
- [Derived] Perou R, Elliott MN, Visser SN, Claussen AH, Scott KG, Beckwith LH, Howard J, Katz LF, Smith DC. Legacy for ChildrenTM: a pair of randomized controlled trials of a public health model to improve developmental outcomes among children in poverty. BMC Public Health. 2012 Aug 23;12:691. doi: 10.1186/1471-2458-12-691. PMID 22917446